CLINICAL TRIAL: NCT01547611
Title: Outcome of Physiotherapy After Surgery for Cervical Disc Disease: a Prospective Randomised Multi-Centre Trial
Brief Title: Outcome of Physiotherapy After Surgery for Cervical Disc Disease: a Prospective Multi-Centre Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: University Hospital, Linkoeping (Other); Karolinska University Hospital (Other); Ryhov County Hospital (Other); Lund University Hospital (Other)
Responsible Party: Principal Investigator, Anneli Peolsson, Assoc. Prof., PhD, MSc PT, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rehab. after cervical surgery
Record Dates: First submitted 2012-02-27; First posted 2012-03-08 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Radiculopathy
Keywords: Rehabilitation; Cervical Spine; Radiculopathy; Disc; Surgery
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Customary treatment (Active Comparator): Group A (physiotherapy as usual), customary treatment. The staff at the Neurosurgical clinic will give the patient ordinary pre- and postoperative information. The physiotherapist at the Neurosurgical clinic informs the patients what to avoid the first weeks after surgery and the importance of a good posture and ergonomic thinking in daily life. The patient is also instructed how to do exercises for the shoulder range of motion. Patients have ordinary post-surgery visit to the surgeon and to the physiotherapist about 6 weeks after the surgery, where physiotherapist instructs the patient in exercises for active neck range of motion.
  Interventions: Other: Customary treatment
- structured behavioural medicine program (Experimental): Group B (extended physiotherapy treatment), customary treatment (please see above) plus a standardised and structured behavioural medicine program. The behavioural medicine program includes functional behavioural analysis of the problem, medical exercise therapy, strategies to increase self-efficacy in activities and problem-solving strategies for coping with disability.
  Interventions: Other: Structured behavioural medicine program

INTERVENTIONS:
Other: Customary treatment — The staff at the Neurosurgical clinic will give the patient ordinary pre- and postoperative information. The physiotherapist at the Neurosurgical clinic informs the patients what to avoid the first weeks after surgery and the importance of a good posture and ergonomic thinking in daily life. The patient is also instructed how to do exercises for the shoulder range of motion. Patients have ordinary post-surgery visit to the surgeon and to the physiotherapist about 6 weeks after the surgery, where physiotherapist instructs the patient in exercises for active neck range of motion.
  Arms: Customary treatment
Other: Structured behavioural medicine program — The behavioural medicine program includes functional behavioural analysis of the problem, medical exercise therapy, strategies to increase self-efficacy in activities and problem-solving strategies for coping with disability.
  Arms: structured behavioural medicine program

SUMMARY:
Many patients with cervical disc disease have long-lasting and complex symptoms with chronic pain, low levels of physical and psychological function and sick-leave. Surgery on a few segmental levels might be expected to solve the disc-specific pain but not the non-specific neck pain and the patients'illness. As much as 2/3 of the patients have been reported to have remaining physical/ psychological disability long-term after surgery. A structured physiotherapy programme after surgery may improve patients'function and return to work. The main purpose of the study is to evaluate what a well structured rehabilitation program adds to the customary treatment after surgery for radiculopathy due to cervical disc disease in respect to function, disability, workability and cost effectiveness. The study is a prospective randomised controlled multi-centre study, with an independent and blinded investigator comparing two alternatives of rehabilitation. 200 patients in working age, with cervical disc disease with clinical findings and symptoms of cervical nerve root compression will be included after informed consent. After inclusion in the study patients will be randomised to one out of the two alternatives of physiotherapy, (A) customary treatment (information/ advice on the specialist clinic) or (A+B) active physiotherapy; standardised and structured program of neck specific exercises combined with a behavioural approach plus customary treatment. Patients will be evaluated both clinically and with questionnaires before surgery, 6 weeks, 3 months, 6 months, 12 months and 24 months after surgery. Main outcome variable are neck specific disability. Cost-effectiveness will be calculated. The inclusion will preliminary be closed 2012. The study could contribute to a better clinical decision making, a better health care which will reduce physical, mental and social costs for the patients, and improve the rates of patients returning to and staying at work.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included from four Neurosurgical clinics in the south of Sweden and the rehabilitation will be performed in primary care units in several counties.
* Patients in working age, with MRI-verified cervical disc disease with clinical findings and symptoms of cervical nerve root compression and who have had surgery with anterior decompression and fusion or posterior surgery (foraminotomy/ laminectomy) will be included after informed consent.

Exclusion Criteria:

* Patients with myelopathy or with a disease or trauma contraindicated to perform the treatment program or the measurements will be excluded and so also patients with lack of familiarity of the Swedish language or with known drug abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2009-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) | Baseline and change after 3, 6, 12 and 24 months follow-up. The outcome measures is going to report a change over time.
  NDI will be measured at baseline before surgical intervention. Change from baseline in NDI will be measured at 3, 6, 12 and 24 months follow-up.
  NDI will be used to investigate Neck specific disability. The 10 sections in the questionnaire are rated on a six-point scale (0-5 point). The scores for all sections are added together and transformed to percentages (where 0% is no pain or difficulties and 100% is highest score for pain and difficulty on all items.

SECONDARY OUTCOMES:
Pain intensity on visual analogue scale (VAS 0-100mm) | The outcome measure is going to report a change over time from baseline and at 6 weeks, 3, 6, 12 and 24 months follow-up
  Pain intensity of neck pain, arm pain and headache, respectively
Dizziness/ unsteadiness measured on a visual analogue scale (VAS) 0-100mm | The outcome measure is going to report a change over time from baseline to 3, 6, 12 and 24 months follow-up
  Dizziness/ unsteadiness measured on a VAS-scale (0=no problems, 100= pretty severe problems).
Modified Odom scale and a question if how important the change is. | The outcome measure is going to report a change over time from before surgery to 6 weeks, 3, 6, 12 and 24 months follow-up.
  A 1 to 6 point scale of treatment outcome. 1=recovered, 2=much better, 3=better, 4=unchanged, 5=worse, 6= much worse. How important is the change on a 0 to 10 point horizontal scale (0=not at all important, 10= very important).
Expectations of treatment fulfilled | The outcome measure is going to report a change from 6 weeks, 3, 6, 12 and 24 months follow-up.
  Fulfillment of the expectations for surgery at follow-ups was measured on a four-grade scale (1=yes, completely; 2=yes, partially; 3=no, not at all; or 4= do not know).
Background data | Mainly before treatment started. Some basic background data are also asked at the follow-ups at 6 weeks, 3, 6, 12 and 24 months to control for variations over time.
  Pain history, pain debute, pain duration, pain medication, other diseases and problems than from the neck, age, sex, smoking, family and social life, expectations of the treatment, care seeking, type of work
Vocational situation | Before intervention and at 3, 6, 12 and 24 months follow-up. The outcome measure is going to report a change over time.
  Questionns about sick-leave, ergonomics, expectations of being able to work in 6 months, work ability index
Pain-drawing | Before intervention and at 3, 6, 12 and 24 months follow-up. The outcome measure is going to report a change over time.
  Character of pain, number of pain localisation and distributions of symptoms
Zung questionnaire | Before intervention and at 3, 6, 12 and 24 months follow-up. The outcome measure is going to report a change over time.
MSPQ questionnaire | Before intervention and at 3, 6, 12 and 24 months follow-up. The outcome measure is going to report a change over time.
Distress and risk assessment method (DRAM) | Before intervention and at 3, 6, 12 and 24 months follow-up. The outcome measure is going to report a change over time.
  Zung and MSPQ questionnaires will be combined in the DRAM instrument
Patient Enablement Instrument (PEI) | Before intervention and at 3, 6, 12 and 24 months follow-up. The outcome measure is going to report a change over time.
Coping Strategies Questionnaire | Before intervention and at 3, 6, 12 and 24 months follow-up. The outcome measure is going to report a change over time.
Work Ability Index | Before intervention and at 6, 12 and 24 months follow-up. The outcome measure is going to report a change over time.
Physical activity/ exercise habits | Before intervention and at 3, 6, 12 and 24 months follow-up. The outcome measure is going to report a change over time.
Symptom satisfaction | Before intervention and at 3, 6, 12 and 24 months follow-up. The outcome measure is going to report a change over time.
  How patients would feel about having their current neck symptoms for the rest of their lives was rated on a seven grade scale (1= delighted, 7=terrible).
Pain frequency and pain medication | Before intervention and at 3, 6, 12 and 24 months follow-up. The outcome measure is going to report a change over time.
Self-efficacy scale | Before intervention and at 3, 6, 12 and 24 months follow-up. The outcome measure is going to report a change over time.
  "People´s beliefs about their capabilities to produce designated levels of performance that exercise influence overe events that affect their lives" Self efficacy (Altmaier) is a 20 item, 11 point scale (0=not at all confident, 10=completely confident).
Question about re-surgery | Before intervention and at 6, 12 and 24 months follow-up. The outcome measure is going to report a change over time.
  Descriptive data
EuroQuol five dimensions self report (EQ-5D) and EuroQuol thermometer | Before intervention and at 3, 6, 12 and 24 months follow-up. The outcome measure is going to report a change over time.
  Health realted quality of life
Multidimensional Pain Inventory, Swedish version (MPI-S), MPI-S significant others and open questions | Before intervention and at 12 and 24 months follow-up. The outcome measure is going to report a change over time.
  Relationship and support from spouses
Neurological status | Before intervention and at 3, 6, 12 and 24 months follow-up. The outcome measure is going to report a change over time.
  Questions of numbness and tinglings in the arm and hand and pain distribution. Clinical examination: sensibility, reflexes, motor function.
Patient Specific Functional Scale (PSFS) | Before intervention and at 3, 6, 12 and 24 months follow-up. The outcome measure is going to report a change over time.
Physical clinical outcome measures | Before intervention and at 3, 6, 12 and 24 months follow-up. The outcome measure is going to report a change over time.
  Range of motion in the neck, head repositioning accuracy (cervical kinesteshia), hand strength, balance (sharpened Romberg, walking in a figure of eight), neck muscle endurance
Patients income | At baseline and at 1 and 2 years follow up. The outcome is going to report a change over time
  Will be used for health echonomic calculations
Copy of the sick-leave receipt from the surgeon | After surgery (baseline, before physiotherapy started)
  Copy of the sickness certificate written by the physician. The certificate will be analysed due to quality with the emphasis on how the cervical radiculopathy impact on function and work ability and due to the quality of sickness certificate in relation to Swedish insurance office rules.

CONTACTS AND LOCATIONS:
Overall Officials: Anneli Peolsson, PhD, Study Chair — Linkoeping University
Locations (2):
- Sweden (2):
  - Department of Medical and Health Sciences, Linköping, Östergötland County
  - Linköping University, Linköping, Östergötland County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peolsson A, Lofgren H, Dedering A, Kristedal M, Oberg B, Zsigmond P, Wibault J. Neurological outcomes after surgery and postoperative rehabilitation for cervical radiculopathy due to disc disease: a 2-year-follow-up of a randomized clinical trial. Sci Rep. 2023 Mar 7;13(1):3830. doi: 10.1038/s41598-023-31005-z. PMID 36882483
- [Derived] Peolsson A, Wibault J, Lofgren H, Dedering A, Oberg B, Zsigmond P, Wahlin C. Work Ability After Anterior Cervical Decompression and Fusion Followed by a Structured Postoperative Rehabilitation: Secondary Outcomes of a Prospective Randomized Controlled Multi-Centre Trial with a 2-year Follow-up. J Occup Rehabil. 2022 Sep;32(3):473-482. doi: 10.1007/s10926-021-10015-6. Epub 2021 Dec 11. PMID 34894316
- [Derived] Lam K, Peolsson A, Soldini E, Lofgren H, Wibault J, Dedering A, Oberg B, Zsigmond P, Barbero M, Falla D. Larger pain extent is associated with greater pain intensity and disability but not with general health status or psychosocial features in patients with cervical radiculopathy. Medicine (Baltimore). 2021 Feb 26;100(8):e23718. doi: 10.1097/MD.0000000000023718. PMID 33663038
- [Derived] Liew BXW, Peolsson A, Falla D, Cleland JA, Scutari M, Kierkegaard M, Dedering A. Mechanisms of recovery after neck-specific or general exercises in patients with cervical radiculopathy. Eur J Pain. 2021 May;25(5):1162-1172. doi: 10.1002/ejp.1741. Epub 2021 Feb 24. PMID 33533164
- [Derived] Liew BXW, Peolsson A, Scutari M, Lofgren H, Wibault J, Dedering A, Oberg B, Zsigmond P, Falla D. Probing the mechanisms underpinning recovery in post-surgical patients with cervical radiculopathy using Bayesian networks. Eur J Pain. 2020 May;24(5):909-920. doi: 10.1002/ejp.1537. Epub 2020 Feb 21. PMID 31985097
- [Derived] Peolsson A, Lofgren H, Dedering A, Oberg B, Zsigmond P, Hedevik H, Wibault J. Postoperative structured rehabilitation in patients undergoing surgery for cervical radiculopathy: a 2-year follow-up of a randomized controlled trial. J Neurosurg Spine. 2019 Mar 22;31(1):60-69. doi: 10.3171/2018.12.SPINE181258. Print 2019 Jul 1. PMID 30901755
- [Derived] Wibault J, Oberg B, Dedering A, Lofgren H, Zsigmond P, Peolsson A. Structured postoperative physiotherapy in patients with cervical radiculopathy: 6-month outcomes of a randomized clinical trial. J Neurosurg Spine. 2018 Jan;28(1):1-9. doi: 10.3171/2017.5.SPINE16736. Epub 2017 Nov 3. PMID 29087809
- [Derived] Peolsson A, Oberg B, Wibault J, Dedering A, Zsigmond P, Bernfort L, Kammerlind AS, Persson LC, Lofgren H. Outcome of physiotherapy after surgery for cervical disc disease: a prospective randomised multi-centre trial. BMC Musculoskelet Disord. 2014 Feb 6;15:34. doi: 10.1186/1471-2474-15-34. PMID 24502414